CLINICAL TRIAL: NCT07251556
Title: Effect of Glucagon-Like Peptide-1 (GLP-1) Receptor Agonists on Subclinical Atherosclerosis in Non-diabetic Patients With Psoriatic Arthritis - a Proof-of-concept Randomized Study
Brief Title: GLP-1 Receptor Agonists in Non-diabetic Patients With Psoriatic Arthritis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho SO, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1
Record Dates: First submitted 2025-09-26; First posted 2025-11-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis Arthritis
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- semaglutide (Experimental): Patients in the treatment group will be started on an initial dose of semaglutide 0.25 mg once weekly for 4 weeks to assess the tolerability of the drug and to minimize potential gastrointestinal side effects. Then 4 weeks the dose will be increased to 0.5 mg once weekly. After 8 weeks the dose will be increased to 1.0mg once weekly for a total treatment period of 24 weeks.
  Interventions: Drug: Semaglutide 0.5 mg; Drug: Semaglutide 1.0 mg; Drug: Semaglutide 0.25 mg
- Control (Other): No active drug administered
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Semaglutide 0.5 mg — Then 4 weeks the dose will be increased to 0.5 mg once weekly.
  Other Names: ozempic
  Arms: semaglutide
Drug: Semaglutide 1.0 mg — 1.0 mg once weekly for 16 weeks
  Other Names: ozempic
  Arms: semaglutide
Drug: Semaglutide 0.25 mg — Initial dose of semaglutide 0.25 mg once weekly for 4 weeks to assess the tolerability of the drug and to minimize potential gastrointestinal side effects.
  Other Names: ozempic
  Arms: semaglutide
Other: No intervention — No intervention
  Arms: Control

SUMMARY:
Background Psoriatic arthritis (PsA) patients are at increased risk of cardiovascular disease. Glucagon-Like Peptide-1 (GLP-1) receptor agonists are cardiovascular protective in diabetics. They have also anti-inflammatory properties. It is hypothesized GLP-1 receptor agonists can prevent the progression of atherosclerosis due to the combination of metabolic factors and disease activity control in non-diabetic PsA patients.

Objectives To investigate the vascular effects of GLP-1 receptor agonists in PsA patients without diabetes. Their metabolic and anti-inflammatory roles will also be examined.

Design and subjects This is a pilot randomized open-labelled trial. We plan to enroll 40 non-diabetic patients with PsA. Participants will be randomized 1:1 to either GLP-1 receptor agonist (semaglutide) or control group.

Study instruments Subclinical carotid artherosclerosis is assessed by high-resolution ultrasound. Arterial stiffness is measured using pulse wave velocity by a tonometry system, and augmentation index by the SphygmoCor device. These assessments will be done at baseline and 24 weeks. Drug adversities will also be documented. Anthropometric measurements, sugar metabolism and lipid levels as well as the PsA disease activity will be monitored.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is associated with an elevated risk of cardiovascular disease (CVD), which contributes to significant morbidity and mortality. A pooled analysis of 11 studies showed that comparing with the general population, there was a 43% higher risk of cardiovascular (CV) event. PsA increases the susceptibility to atherosclerosis through chronic inflammation, high prevalence of traditional CV risk factors, and the impact of medications. Therefore, there is a possibility that suppression of underlying inflammation, combined with effective control of CV risk factors, could potentially disrupt the accelerated development of atherosclerosis and subsequently improve the CV outcomes of patients with PsA.

Glucagon-like peptide-1 receptor agonists (GLP-1) receptor agonists are a new class of antidiabetic medications. Their beneficial effects on CV endpoints in diabetes mellitus (DM) are well-proven. GLP-1 receptor agonists were also reported to reduce the progression of carotid intima-media thickness (CIMT) independently of its effect on glucose control after 8 months in patients with DM. However, their effects on CV outcomes in patients with non-DM remain uncertain. The initial SCALE group of trials studied GLP-1 receptor agonists in non-diabetic patients with higher body mass index (BMI) and found promising results in terms of reducing body weight, blood pressure, and hemoglobin A1c (HbA1c). The SELECT study, a recent landmark large randomized controlled trial, revealed the addition of semaglutide, a long-acting analogue of GLP-1, to standard care was superior to placebo in reducing the risk of major adverse CV events among overweight patients with preexisting CVD who were non-diabetic.

On top of being CV protective, the potential anti-inflammatory properties of GLP-1 receptor agonists make them appealing treatment option for patients with inflammatory arthritis. GLP-1 receptor agonists inhibit lipopolysaccharide-induced inflammation by phosphorylating AMP-activated protein kinase, which leads to the inhibition of the nuclear factor kappa B (NF-κB) pathway. This inhibition is associated with a decrease in the expression of proinflammatory genes responsible for producing various cytokines such as tumor necrosis factor-α and Interleukin-6 that play important roles in the pathogenesis of arthritis. Additionally, GLP-1 receptor agonists have been found to prevent phosphorylation of IκBα, a key inhibitory protein that normally prevents nuclear translocation of NF-κB transcription factors responsible for downstream proinflammatory cytokine production.

Obesity is a pro-inflammatory state which is prevalent in PsA. Weight loss is associated with improved disease activity in PsO and PsA. A recent meta-analysis showed that compared with the control group, lifestyle interventions involving weight loss significantly improved the mean change of Psoriasis Area and Severity Index (PASI) in psoriasis. The CV protective and therapeutic effects of GLP-1 receptor agonists in PsA have not been studied. There is a small observational study involving patients with rheumatoid arthritis (RA) (n=11) and PsA (n=4), which showed an improvement after GLP-1 receptor agonists treatment in disease activity score 28-joint from 4.2 to 2.7 among the responders.

Carotid ultrasound is a noninvasive imaging technique that can identify the presence of carotid plaque and increased CIMT, representing an unequivocal manifestation of atherosclerosis and serving as a surrogate for CVD. We have shown that subclinical carotid atherosclerosis (SCA) was more prevalent in PsA than controls, even without CV risk factors. In PsA, the presence of SCA is linked to a higher risk of future CV events. Moreover, arterial stiffness also serves as a surrogate marker for CV risk. Each 1.0 m/s increase in brachial-ankle pulse wave velocity (ba-PWV) was reported to associate with a 12% rise in the occurrence of total CV events after adjusting for traditional risk factors.

In light of the potential multitude anti-atherosclerosis effects of GLP-1 receptor agonists, we would like to conduct the first interventional study evaluating the efficacy of semaglutide as disease modifying therapy in atherosclerosis in non-diabetic patients with PsA. Two established surrogate markers for CVD will be used. The results of the study will contribute preliminary data and mechanistic insights regarding the possible effects of GLP-1 receptor agonists on arterial wall, atherosclerotic plaques, and PsA disease activity. Promising results will prompt a properly designed study with adequate power to assess the multidimensional efficacy of GLP-1 receptor agonists in patients with PsA that could reshape the future management of PsA patients in terms of CV risk prevention.

ELIGIBILITY:
Inclusion Criteria:

1. fulfill the ClASsification criteria for Psoriatic Arthritis,
2. are rheumatoid factor negative,
3. BMI >=25 kg/m2,
4. are over 18 years old and
5. Chinese subjects

Exclusion Criteria:

1. have prior therapy with GLP-1 receptor agonists during the last 24 weeks,
2. have pre-existing diabetes,
3. have liver or renal impairment,
4. have known or symptoms suggestive of CVD,
5. have chronic or previous acute pancreatitis,
6. have current malignancy,
7. are pregnant, breastfeeding or of childbearing potential, or
8. are unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the proportion of subjects with CIMT between the semaglutide group and control group over a period of 24 weeks. | 24 weeks
  carotid artery intima media thickness by ultrasound

SECONDARY OUTCOMES:
Carotid plaque progression | 24 weeks
  Plaque progression is defined as an incident plaque in a segment without plaque before or an increase in number of plaque.
total plaque area (TPA) | 24 weeks
  For TPA, the plane for measurement of each plaque will be chosen by reviewing the video of the scan to find the largest extent of plaque as seen on the longitudinal view.
BMI | 24 weeks
  weight in kilograms/the square of height in meters
waist circumferences | 24 weeks
  in centimeters
sugar profile | 24 weeks
  Fasting blood glucose
sugar profile | 24 weeks
  HbA1c
lipid profile | 24 weeks
  low-density lipoprotein-cholesterol
lipid profile | 24 weeks
  triglycerides
Occurrence of adverse events. | 24 weeks
  The treating physicians will record all adverse events and serious adverse events
PsA disease activity (MDA) | 24 weeks
  Percentage of patients in MDA, a composite of number of swollen joints (0-66), number of tender joints (0-68), visual analogue scale (VAS, score in 0-10) for pain, VAS for patient's global assessment, the Leeds Enthesitis Index, PASI and Health Assessment Questionnaire Disability Index
PsA disease activity (DAPSA) | 24 weeks
  A composite of C-reactive protein, swollen joint count, tender joint count, patient pain VAS and patient global VAS